CLINICAL TRIAL: NCT07256691
Title: Effect of Calcium-Based Bioceramic Sealer and Resin-Based Sealer on Postoperative Pain in Adults With Asymptomatic Apical Periodontitis
Brief Title: Effect of Calcium-Based Bioceramic Sealer and Resin-Based Sealer on Postoperative Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fatima Memorial Hospital (Other)
Responsible Party: Principal Investigator, SHEHRYAR KHAN, Principal investigator, Fatima Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMH-13/06/2025-IRB-1673
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Asymptomatic Apical Periodontitis
Keywords: Bioceramic sealer; Resin-based sealer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: This is a double-blind study where both the participant and the care provider (dentist performing the root canal treatment) are blinded to the type of sealer used. Additionally, the outcome assessor (person recording postoperative pain levels) is also blinded to the sealer material used. The sealers are coded and labeled in a way that prevents both the provider and participant from identifying which material is being used during the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bioceramic Sealer Group (Experimental): Patients in this group will receive root canal obturation using bioceramic (calcium silicate-based) sealer with gutta-percha. Postoperative pain will be assessed at 4, 24, and 48 hours using the Numeric Pain Rating Scale (NPRS).
  Interventions: Procedure: Bioceramic sealer obturation
- Resin-Based Sealer Group (Experimental): Patients in this group will receive root canal obturation using resin-based sealer with gutta-percha. Postoperative pain will be assessed at 4, 24, and 48 hours using the Numeric Pain Rating Scale (NPRS).
  Interventions: Procedure: Resin-based sealer obturation technique

INTERVENTIONS:
Procedure: Resin-based sealer obturation technique — Root canal obturation using resin based sealer with single cone GP technique. Canals prepared and irrigated as above. Pain recorded at 4, 24, and 48 hours post-obturation using NPRS.
  Arms: Resin-Based Sealer Group
Procedure: Bioceramic sealer obturation — Participants in this group will undergo root canal obturation using a calcium silicate based bioceramic sealer with a single-cone gutta percha technique. After standard canal preparation and irrigation with 2.5% sodium hypochlorite, the canals will be dried with paper points. The bioceramic sealer will be applied using a lentulospiral or directly coated on the master gutta-percha cone. A matched-taper gutta-percha cone will then be inserted to full working length. The canal orifice will be sealed with a temporary or permanent restoration. Postoperative pain will be assessed at 4, 24, and 48 hours using the Numeric Pain Rating Scale (NPRS).
  Arms: Bioceramic Sealer Group

SUMMARY:
This study aims to compare the effect of calcium-based bioceramic sealer and resin-based sealer on postoperative pain in adult patients with asymptomatic apical periodontitis undergoing root canal treatment. Asymptomatic apical periodontitis is a condition where the tissue around the tip of the tooth root is inflamed or shows a lesion on X-ray, but the patient does not experience pain.

A total of 60 patients will be randomly assigned to receive root canal treatment with either the bioceramic sealer (Group A) or the resin-based sealer (Group B). Pain after treatment will be measured using a 0-10 Numeric Pain Rating Scale at 4, 24, and 48 hours post-treatment. The highest pain score reported will determine whether the treatment is considered a success (no or mild/moderate pain) or failure (severe pain).

The results of this study will provide evidence on which sealer is associated with less postoperative pain, helping clinicians make informed decisions about root canal filling materials.

DETAILED DESCRIPTION:
This randomized controlled clinical trial aims to compare calcium-based bioceramic sealer and resin-based sealer in root canal treatment for adult patients with asymptomatic apical periodontitis. Asymptomatic apical periodontitis is a condition where the tissue around the tip of the tooth root is inflamed or shows a lesion on X-ray, but the patient does not feel pain.

A total of 60 patients aged 18-55 years will be recruited at the Department of Operative Dentistry, Fatima Memorial Hospital, Lahore. Eligible patients will have non-vital teeth with fully formed roots and periapical lesions classified as PAI scores 2-4. Patients with systemic diseases, periodontally compromised teeth, or complications during treatment will be excluded.

Patients will be randomly assigned to two groups: Group A will receive root canal obturation using bioceramic sealer, and Group B will receive resin-based sealer. The treatment procedure involves standard root canal cleaning and shaping, irrigation, and obturation using a single-cone technique with Gutta-percha.

Postoperative pain will be assessed using a Numeric Pain Rating Scale (0-10) at 4, 24, and 48 hours after obturation. The highest pain score reported across these time points will determine the outcome. Pain levels will be classified as: None (0), Mild (1-3), Moderate (4-7), or Severe (8-10). Patients with severe pain (8-10) will be considered treatment failures, while all others will be considered treatment successes.

Data will be analyzed using SPSS. Descriptive statistics will summarize demographic and clinical variables, and Chi-square tests will compare postoperative pain between groups. The study aims to provide evidence on which sealer results in less postoperative pain, supporting better clinical decision-making in endodontics.

ELIGIBILITY:
Inclusion Criteria:Age 18-55 years.

* Both genders.
* Teeth diagnosed with asymptomatic apical periodontitis.
* Teeth are asymptomatic (no pain on percussion or palpation).
* Non-vital pulp (no response on Electric Pulp Testing).
* Teeth with fully formed apices.
* Teeth with Periapical Index (PAI) scores 2-4 on radiographs.

Exclusion Criteria:

* Medically compromised patients (e.g., those with immunosuppressive or systemic diseases, or on medications that may affect healing).
* Patients who refuse to participate or are unable to communicate their symptoms (e.g., due to psychological disorders).
* Teeth where full working length cannot be reached.
* Periodontally compromised teeth (probing depth >4 mm).
* Complications during treatment (e.g., separation of a file, ledging).
* Overfilling (filling beyond the radiographic apex) or short filling (>2 mm from the radiographic apex).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 4, 24, and 48 hours after root canal obturation.
  Pain intensity will be measured using the Numeric Pain Rating Scale (0-10). The highest score among the three time points will determine outcome. Scores 0-7 are considered successful; 8-10 indicate failure.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatima Memorial Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The IPD shared will include demographic information, clinical findings, pain scores, and treatment details for each patient.